CLINICAL TRIAL: NCT03613207
Title: An Exploratory Pilot Study in Healthy Volunteers to Assess the Parameters for the Design of Bioequivalence Studies on Moderately Lipophilic, Moderately to Highly Protein Bound Drugs Using Dermal Open Flow Microperfusion (dOFM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joanneum Research Forschungsgesellschaft mbH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDA02_AIM2_PILOT; DRKS00012706 (Registry Identifier: German Clinical Trials Register)
Record Dates: First submitted 2018-07-03; First posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-07

CONDITIONS: Dermatology/Skin - Other; Dermal Pharmacokinetic Measurements
Keywords: Dermal open flow microperfusion; dOFM
MeSH Terms: interventions — Lidocaine; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dermal pharmacokinetic measurement (Experimental): Measurement of dermal pharmacokinetic (PK) parameters (AUC, Cmax) within each subject.
  For dermal PK measurement cutaneous interstitial fluid will be sampled using dermal open flow microperfusion (dOFM). Additionally 8 blood samples will be drawn to rule out systemic appearance of lidocaine/prilocaine.
  Each subject will have 9 test sites in total which are treated with:
  * 2 test sites: 15 mg/cm² lidocaine and prilocaine cream (2.5% lidocaine, 2.5% prilocaine, ACTAVIS LABORATORIES UT INC, US)
  * 2 test sites: 10 mg/cm² lidocaine and prilocaine cream (2.5% lidocaine, 2.5% prilocaine, ACTAVIS LABORATORIES UT INC, US)
  * 2 test sites: 5 mg/cm² lidocaine and prilocaine cream (2.5% lidocaine, 2.5% prilocaine, ACTAVIS LABORATORIES UT INC, US)
  * test sites: 10 mg/cm² Oraqix® gel (2.5% lidocaine, 2.5% prilocaine, Dentsply Pharmaceutical Inc., US/Dentsply DETRY GmbH, Germany)
  * 2 test sites: untreated test site
  Interventions: Other: Dermal pharmacokinetic measurement; Drug: Lidocaine and prilocaine cream; Drug: Oraqix® gel; Device: dOFM-System; Procedure: Blood sampling

INTERVENTIONS:
Other: Dermal pharmacokinetic measurement — * Each subject will have 9 test sites: 4 on the left thigh, 4 on the right thigh, 1 on the arm
  * Each test site receives 2 dOFM probes
  * Dosing:
    * 2 test sites: 15 mg/cm² lidocaine and prilocaine cream (2.5% lidocaine, 2.5% prilocaine, ACTAVIS LABORATORIES UT INC, US)
    * 2 test sites: 10 mg/cm² lidocaine and prilocaine cream (2.5% lidocaine, 2.5% prilocaine, ACTAVIS LABORATORIES UT INC, US)
    * 2 test sites: 5 mg/cm² lidocaine and prilocaine cream (2.5% lidocaine, 2.5% prilocaine, ACTAVIS LABORATORIES UT INC, US)
    * 1 test site: 10 mg/cm² Oraqix® gel (2.5% lidocaine, 2.5% prilocaine, Dentsply Pharmaceutical Inc., US/Dentsply DETRY GmbH, Germany)
    * 2 test sites: untreated test site
  * ISF sampling: 24 hours post-dose
  * Blood sampling: 7 samples post-dose
Drug: Lidocaine and prilocaine cream — lidocaine and prilocaine cream (2.5% lidocaine, 2.5% prilocaine, ACTAVIS LABORATORIES UT INC, US) will be applied to 6 test sites per subject
Drug: Oraqix® gel — Oraqix® gel (2.5% lidocaine, 2.5% prilocaine, Dentsply Pharmaceutical Inc., US/Dentsply DETRY GmbH, Germany) will be applied to 1 test site per subject
Device: dOFM-System — Dermal open flow microperfusion system will be used to collect interstitial fluid in order to assess lidocaine/prilocaine concentrations over 24 hours
Procedure: Blood sampling — 8 blood samples will be collected in order to assess systemic lidocaine/prilocaine concentrations pre-dose (1 sample) and 24 hours post dose (7 samples)

SUMMARY:
The overall aim of this clinical pilot study is to develop an optimal design (e.g. dose, study duration) for the main clinical study. In the main study factors that influence dOFM data variability will be measured to develop a general BE testing method using dOFM for dermatological drug products.

DETAILED DESCRIPTION:
In this herein described pilot study 6 subjects will receive three different topical doses of Lidocaine 2.5% and Prilocaine 2.5% cream (2.5% lidocaine, 2.5% prilocaine, ACTAVIS LABORATORIES UT INC, US ) to select an optimal dose for the main study. Oraqix® gel (2.5% lidocaine, 2.5% prilocaine, Dentsply Pharmaceutical Inc., US) will be applied to assess whether it can be used as negative control in the main study. Blood samples will also be drawn at prior to dosing to establish a baseline, and at defined time points post-dose to assess systemic drug levels. Furthermore, lateral diffusion from a dosed site to an adjacent (non-dosed) test site will be evaluated in this pilot study. Different non-invasive devices will be tested to identify influencing factors for skin penetration in order to complete the available information on skin characteristics for the main study.

This pilot will be a single center, open label, exploratory research study to assess the dermal PK of marketed topical formulations of lidocaine/prilocaine in six healthy volunteers using dOFM. The study will be performed at the Clinical Research Center of the Medical University of Graz/Austria.The study comprises three visits, a screening visit (Visit 1), a study visit of approximately 28 h (Visit 2) for application of dermatological drug products, and an End-of-Study visit (Visit 3). In Visit 2 each subject will have nine test sites, four on the left thigh, four on the right thigh (resulting in 8 test sites on both thighs) and one on the arm. Each of the nine test site will have 2 dOFM probes resulting in 18 dOFM probes per subject. On six of the eight test sites on the thighs three different doses of Lidocaine 2.5% and Prilocaine 2.5% cream cream will be applied (5 mg/cm², 10 mg/cm² or 15 mg/cm²) to assess the dose for the main study. On another test site on the thighs Oraqix® gel will be applied to check if Oraqix® can be used as negative control in the main study. On the remaining test site on the thighs as well as on the test site on the arm no products will be applied to test for potential cross-talk between test sites by lateral diffusion and systemic redistribution, resulting in seven treated and two non-treated sites per subject. Additionally 8 blood samples will be drawn to rule out systemic appearance of lidocaine and/or prilocaine. Further, devices to identify possible factors influencing skin penetration will be measured on each thigh (e.g. TEWL).

ELIGIBILITY:
Inclusion Criteria:

Subject candidates must fulfill all of the following inclusion criteria to be eligible for participation in the study, unless otherwise specified:

1. 18 to 65 years inclusive,
2. Males and/or non-pregnant, non-breastfeeding females (subjects need to be informed about adequate contraceptive methods).
3. Able to read, understand, and sign the written informed consent form.
4. Willing to follow the protocol requirements and comply with protocol restrictions.

Exclusion Criteria:

Subject candidates must not be enrolled in the study if they meet any of the following criteria:

1. Social Habits

   1. Smoker who is not willing to restrain from smoking during the in-house-visit (Visit 2).
   2. History of drug and/or alcohol abuse within one year of start of study as judged by the investigator.
2. Medications

   a. Use of any medications (specially medication referred in the prescription information of the products) other than hormonal contraceptive or hormone replacement therapy within the 7 days or 5 half-life periods whichever is longer prior to the initial dose of study medication.
3. Diseases

   1. Congenital or idiopathic methemoglobinemia
   2. Glucose-6-phosphate dehydrogenase deficiencies
   3. Presence of any acute or chronic disease or malignancies unless deemed not clinically significant by the investigator.
4. Any reason which, in the opinion of the investigator, would prevent the subject from safely participating in the study.
5. Any abnormalities found at physical examination or vital signs, unless deemed not clinically significant by the investigator.
6. Clinically significant abnormal laboratory evaluation results, as deemed by the investigator.
7. Clinically significant abnormal 12-lead ECG at screening, as deemed by the investigator.
8. Positive results to the test for Hepatitis B antigen or Hepatitis C antibodies.
9. Positive HIV test.
10. Positive alcohol breath test.
11. Blood donation within 30 days or significant loss of blood or plasma (more than 550 ml) within 90 days prior to screening.
12. Subjects who have received an investigational drug within 30 days prior to the initial dose of study medication.
13. Any food allergy, intolerance, restriction or special diet that, in the opinion of the investigator, could contraindicate the subject's participation in this study.
14. Known or suspected allergy/hypersensitivity to lidocaine or prilocaine, known history of sensitivity to local anesthetics of the amide type or to any other component of the product, other related products, or any inactive ingredients.
15. Tattoos or broken and/or damaged skin at the application areas.
16. Active skin diseases like psoriasis or atopic dermatitis judged by the investigator.
17. Scarring at the anterior part of the thighs
18. Subjects prone to keloid or hypertrophic scar formation or any known wound healing disorder.
19. Recent and/or recurrent history of autonomic dysfunction (e.g., recurrent episodes of fainting, palpitations, etc.) judged by the investigator.
20. Not willing to avoid excessive sun exposure, steam baths, sauna, swimming and other strenuous activities between Visit 2 and the End-of-Study examination to ensure good tissue regeneration.
21. Not willing to refrain from shaving the anterior of the thighs or using skin care products on the anterior of the thighs for at least 5 days prior to start of Visit 2.
22. Pronounced hairiness on the thighs that may negatively affect BE testing.
23. Known allergy/hypersensitivity to any of the materials/supplies used during the study.
24. Presence of needle phobia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2018-05-03 (Actual)

PRIMARY OUTCOMES:
Find the dose of Lidocaine 2.5% and Prilocaine 2.5% cream for the main study by comparing the concentration time curves and corresponding PK parameter Cmax of 3 different doses (5 mg/cm², 10 mg/cm² and 15 mg/cm²) twice in each subject | 24 hours
  Three different doses (5 mg/cm², 10 mg/cm² and 15 mg/cm²) of Lidocaine 2.5% and Prilocaine 2.5% cream will be dosed twice in each subject in parallel.
  The concentration time curves and the PK parameter Cmax of this three doses will be compared and based on this data the team will decide in collaboration with the FDA project officer which dose will be used for the main study. Thereby study duration and sampling intervals (resolution) for the main study will be defined.
Find the dose of Lidocaine 2.5% and Prilocaine 2.5% cream for the main study by comparing the concentration time curves and corresponding PK parameter AUC of 3 different doses (5 mg/cm², 10 mg/cm² and 15 mg/cm²) twice in each subject | 24 hours
  Three different doses (5 mg/cm², 10 mg/cm² and 15 mg/cm²) of Lidocaine 2.5% and Prilocaine 2.5% cream will be dosed twice in each subject in parallel.
  The concentration time curves and the PK parameter AUC of this three doses will be compared and based on this data the team will decide in collaboration with the FDA project officer which dose will be used for the main study. Thereby study duration and sampling intervals (resolution) for the main study will be defined.

SECONDARY OUTCOMES:
Test for systemic exposure and systemic cross-talk by measuring lidocaine/prilocaine concentrations (µg/ml) in blood samples and ISF samples from a distant untreated test site on the arm | 24 hours
  To measure the degree to which lidocaine and/or prilocaine are absorbed into the skin and are redistributed via the blood stream.
  Lidocaine and Prilocaine concentrations will be measured in blood samples and ISF samples from a distant untreated test site on the arm. If no significant drug concentration are found in the blood samples and in the skin of the untreated topical test site on the arm (relative to the drug concentration of the treated sites) systemic exposure can be excluded.
Test for lateral diffusion (crosstalk between adjacent test sites) by measuring lidocaine/prilocaine concentrations (µg/ml) of untreated test sites | 24 hours
  In one central control site, located between two test sites dosed with lidocaine and prilocaine cream, no drug product will be applied. This setup allows testing for lateral diffusion in the skin. If no significant lidocaine or prilocaine concentration (relative to the drug concentration of the treated sites) in combination with the results from outcome 2 can be found in this untreated test site, lateral diffusion can be excluded.
Check if Oraqix® gel can be used as 'negative control' for bioequivalence testing in the main study by comparing Oraqix® gel with Lidocaine and prilocaine cream (AUC). | 24 hours
  On one test site Oraqix® gel will be applied with a dose of 10 mg/cm² and on another test site lidocain and prilocaine crem will be applied with a dose of 10 mg/cm².
  Oraqix® gel will be compared with lidocaine and prilocaine cream by performing the average bioequivalence test. In accordance with the CDER-Guidance on "Statistical approaches on establishing bioequivalence", the 90% confidence interval for the mean difference of the AUC values will be calculated. Oraqix® gel can be used as 'negative control' if the calculated confidence interval dose not fall within the limits of 0.80 - 1.25.
Check if Oraqix® gel can be used as 'negative control' for bioequivalence testing in the main study by comparing Oraqix® gel with Lidocaine and prilocaine cream (Cmax). | 24 hours
  On one test site Oraqix® gel will be applied with a dose of 10 mg/cm² and on another test site lidocain and prilocaine crem will be applied with a dose of 10 mg/cm².
  Oraqix® gel will be compared with lidocaine and prilocaine cream by performing the average bioequivalence test. In accordance with the CDER-Guidance on "Statistical approaches on establishing bioequivalence", the 90% confidence interval for the mean difference of the Cmax values will be calculated. Oraqix® gel can be used as 'negative control' if the calculated confidence interval dose not fall within the limits of 0.80 - 1.25.

OTHER OUTCOMES:
Skin temperature [°C] | Timepoint -3 hours (pre-dose) and timepoint 23 hours (post-dose)
  Different non-invasive devices will be tested to identify influencing factors for skin penetration in order to complete the available information on skin characteristics for the main study.
TEWL (trans-epidermal water loss) [g/(m²*h)] | Timepoint -3 hours (pre-dose) and timepoint 23 hours (post-dose)
  Different non-invasive devices will be tested to identify influencing factors for skin penetration in order to complete the available information on skin characteristics for the main study.
Skin impedance [Ω];[S];[°] | Timepoint -3 hours (pre-dose) and timepoint 23 hours (post-dose)
  Different non-invasive devices will be tested to identify influencing factors for skin penetration in order to complete the available information on skin characteristics for the main study.
Hair follicle density [n/cm²] | Timepoint -3 hours (pre-dose) and timepoint 23 hours (post-dose)
  Different non-invasive devices will be tested to identify influencing factors for skin penetration in order to complete the available information on skin characteristics for the main study.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pieber, Prof., Principal Investigator — Medical University of Graz
Locations (1):
- HEALTH - Joanneum Research, Graz, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bodenlenz M, Tiffner KI, Raml R, Augustin T, Dragatin C, Birngruber T, Schimek D, Schwagerle G, Pieber TR, Raney SG, Kanfer I, Sinner F. Open Flow Microperfusion as a Dermal Pharmacokinetic Approach to Evaluate Topical Bioequivalence. Clin Pharmacokinet. 2017 Jan;56(1):91-98. doi: 10.1007/s40262-016-0442-z. PMID 27539717
- [Background] Bodenlenz M, Dragatin C, Liebenberger L, Tschapeller B, Boulgaropoulos B, Augustin T, Raml R, Gatschelhofer C, Wagner N, Benkali K, Rony F, Pieber T, Sinner F. Kinetics of Clobetasol-17-Propionate in Psoriatic Lesional and Non-Lesional Skin Assessed by Dermal Open Flow Microperfusion with Time and Space Resolution. Pharm Res. 2016 Sep;33(9):2229-38. doi: 10.1007/s11095-016-1960-y. Epub 2016 Jun 6. PMID 27271272
- [Background] Bodenlenz M, Aigner B, Dragatin C, Liebenberger L, Zahiragic S, Hofferer C, Birngruber T, Priedl J, Feichtner F, Schaupp L, Korsatko S, Ratzer M, Magnes C, Pieber TR, Sinner F. Clinical applicability of dOFM devices for dermal sampling. Skin Res Technol. 2013 Nov;19(4):474-83. doi: 10.1111/srt.12071. Epub 2013 Apr 13. PMID 23581539
- [Background] Dragatin C, Polus F, Bodenlenz M, Calonder C, Aigner B, Tiffner KI, Mader JK, Ratzer M, Woessner R, Pieber TR, Cheng Y, Loesche C, Sinner F, Bruin G. Secukinumab distributes into dermal interstitial fluid of psoriasis patients as demonstrated by open flow microperfusion. Exp Dermatol. 2016 Feb;25(2):157-9. doi: 10.1111/exd.12863. Epub 2015 Nov 23. No abstract available. PMID 26439798
- [Background] Tiffner K, Boulgaropoulos B, Hofferer C, Birngruber T, Porksen N, Linnebjerg H, Garhyan P, Lam ECQ, Knadler MP, Pieber TR, Sinner F. Quantification of Basal Insulin Peglispro and Human Insulin in Adipose Tissue Interstitial Fluid by Open-Flow Microperfusion. Diabetes Technol Ther. 2017 May;19(5):305-314. doi: 10.1089/dia.2016.0384. Epub 2017 Mar 22. PMID 28328234
- See also: n Vivo Dermal Open Flow Microperfusion: A Novel Approach to Evaluating Topical Bioavailability and Bioequivalence — https://www.fda.gov/downloads/Drugs/NewsEvents/UCM591892.pdf